CLINICAL TRIAL: NCT01556490
Title: A Phase III Clinical Trial of Intra-arterial TheraSphere® in the Treatment of Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Efficacy Evaluation of TheraSphere in Patients With Inoperable Liver Cancer
Acronym: STOP-HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS-103
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-08

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Standard-of-care sorafenib, with no added therapy
- Treatment group (Experimental): Standard-of-care sorafenib plus TheraSphere
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — Yttrium 90 microspheres
  Arms: Treatment group

SUMMARY:
The safety and effectiveness of TheraSphere will be evaluated in patients with unresectable hepatocellular carcinoma in whom treatment with standard-of-care sorafenib is planned. All patients receive the standard-of-care sorafenib with or without the addition of TheraSphere.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-related evaluation
* Male or female patients over 18 years of age
* Unresectable HCC confirmed by histology or by non-invasive AASLD criteria
* Measurable disease defined as at least one uni-dimensional measurable lesion by CT or MRI according to RECIST 1.1
* Child Pugh score ≤ 7 points
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤ 1
* Life expectancy of 12 weeks or more
* Eligible to receive standard-of-care sorafenib
* Platelet count of > 50 x 10⁹/L or > 50% prothrombin activity
* Hemoglobin ≥ 8.5 g/dL
* Bilirubin ≤ 2.5 mg/dL
* Alanine transaminase (ALT) and Aspartate Aminotransferase (AST)< 5 X upper limit of normal
* Amylase or lipase ≤ 2X upper limit of normal
* Serum creatinine ≤ 1.5 X upper limit of normal
* International normalized ratio (INR) < 2.0

Exclusion Criteria:

* Main portal vein thrombosis
* Eligible for curative treatment (ablation or transplantation)
* History of previous or concurrent cancer other than HCC unless treated curatively 5 or more years prior to entry
* Confirmed presence of extra-hepatic disease except lung nodules and mesenteric or portal lymph nodes ≤ 2.0 cm each
* Risk of hepatic or renal failure
* Tumor replacement ≥ 70% of total liver volume based on visual estimation by investigator OR tumor replacement ≥ 50% of total liver volume in the presence of albumin <3 mg/dL
* History of severe allergy or intolerance to contrast agents, narcotics sedatives or atropine that cannot be managed medically
* Contraindications to angiography and selective visceral catheterization.
* History of organ allograft
* Known contraindications to sorafenib including allergic reaction, pill-swallowing difficulty, evidence of severe or systemic diseases, uncontrolled severe hypertension or history of cardiac arrhythmias, congestive heart failure . New York Heart Association class 2, myocardial infarct within 6 months, prolonged QT/QTc >450ms, evidence of torsades de pointe, or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial, significant GI bleed within 30 days, metastatic brain disease, renal failure requiring dialysis
* Taking any of the following: Rifampicin, St. John's Wort, phenytoin, carbamazepine, phenobarbital, dexamethasone
* Taking any other systemic anticancer agent (docetaxel, doxorubicin, irinotecan)
* Taking any substrate agents for Cytochrome P450 (CYP) 2B6 (bupropion, cyclophosphamide, efavirenz, ifosfamide, methadone, paclitaxel, amodiaquine, repaglinide)
* Taking any UDP-glucuronosyltransferase (UGT) 1A1 and UGT 1A9 substrates (e.g. irinotecan)
* Taking P-Gp substrates (e.g. Digoxin)
* Prior liver resection must have taken ≥2 months prior to randomization
* Treatment with other locoregional therapies (other than study treatment) has not been planned for the duration of the clinical study period
* Prior external beam radiation treatment to the chest, liver or abdomen
* Prior yttrium-90 microsphere treatment to the liver
* Prior treatment with transarterial chemoembolization (TACE) or bland embolization must have occurred >2 months prior to randomization and must have been applied to a treatment field and/or lobe not targeted for treatment under this protocol. For patients with tumor progression in the treatment field and /or lobe previously treated with TACE, vessels feeding the tumor(s) must be assessed for adequate blood flow using angiography (cone beam computerized tomography (CBCT) strongly recommended), and TACE or bland embolization must have been applied >6 months prior to randomization.
* Anti-cancer therapy or any treatment with an investigational agent within 30 days prior to randomization
* Adverse effects due to prior therapy unresolved at randomization
* Prior systemic treatment for the treatment of HCC, including sorafenib given for more than 4 weeks during the 2 previous months prior to randomization, no prior sorafenib related toxicity
* Evidence of pulmonary insufficiency or inadequately treated moderate grade or severe/very severe grade chronic obstructive pulmonary disease
* Intervention for, or compromise of, the Ampulla of Vater
* Clinically evident ascites (trace ascites on imaging is acceptable)
* Pregnancy or breast feeding
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to randomization
* Disease or condition that would preclude safe use of TheraSphere, including concurrent dialysis treatment, or unresolved serious infections. Patients infected with HIV can be considered, however, they must be well managed and well controlled with undetectable viral load
* Participation in concurrent clinical trials evaluating treatment intervention(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, MBA, Principal Investigator — Dept of Radiology Northwestern University
Locations (93):
- United States (20):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Northshore Hospital, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Wayne State Harper Hospital, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Miami Valley Hospital, Dayton, Ohio
  - Legacy Meridian Park Medical Center, Tualatin, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St Marks Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentra Norfolk General Hospital, Norfolk, Virginia
  - Seattle Cancer Care Alliance/University of Washington Medical Center, Seattle, Washington
- Belgium (2):
  - CUB Hôpital Erasme, Brussels
  - CHU Liege, Liège
- Canada (5):
  - University of Alberta Hspital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre / Royal Victoria Hospital, Montreal, Quebec
  - CHUM St. Luc, Montreal
- France (21):
  - Hôpital Jean Verdier, Bondy
  - CHU Estaing, Clermont-Ferrand
  - APHP Hôpital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU de Grenoble, La Tronche
  - CHU Lyon - Hopital de la Croix Rousse, Lyon
  - Centre Léon-Bérard, Lyon
  - Hopital de la Timone CHU, Marseille
  - Hôpital Saint Eloi, Montpellier
  - CHU Hôtel-Dieu, Nantes
  - CHU de Nice, Nice
  - Hôpital Haut-Lévêque, CHU Bordeaux, Pessac
  - CHU de Poitiers, Poitiers
  - CHU Reims, Reims
  - Centre Eugene Marquis, Rennes
  - CHU Amiens Picardie - Hôpital Sud, Salouël
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Purpan, Toulouse
  - CHU Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
  - Hôpital Universitaire Paul Brousse, Villejuif
- Germany (5):
  - Universitätsklinikum Bonn, Bonn
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig, Klinik für Diagnostische und Interventionelle Radiologie, Leipzig
  - Universitätsklinikum Tübingen, Diagnostische und Interventionelle Radiologie, Tübingen
- Azienda Ospedaliero -Universitaria di Bologna, Bologna, Italy
- Netherlands (6):
  - VUMC, Amsterdam
  - AMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - MUMC, Maastricht
  - Erasmus MC, Rotterdam
- National University Hospital, Singapore, Singapore
- South Korea (5):
  - St. Mary Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (16):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - UDIAT Corporacio Parc Tauli, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Servicio de Radiología, Hospital Universitario Virgen de la Arrixaca., Murcia
  - Hosptal Universitario Central de Asturias (nuevo HUCA), Oviedo
  - Hospital Clínico Universitario, Salamanca
  - H. Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (11):
  - New Queen Elizabeth Hospital Birmingham, Birmingham
  - Addenbrooks Hospital, Cambridge
  - Edinburgh Cancer Centre, Edinburgh
  - Royal Surrey Country Hospital, Guildford
  - Royal Liverpool University Hospital, Liverpool
  - University College London Cancer Institute, London
  - King's College Hospital;, London
  - Imperial College London, London
  - Christie Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Weston Park Hospital, Sheffield, Sheffield

REFERENCES:
- [Derived] Chauhan N, Bukovcan J, Boucher E, Cosgrove D, Edeline J, Hamilton B, Kulik L, Master F, Salem R. Intra-Arterial TheraSphere Yttrium-90 Glass Microspheres in the Treatment of Patients With Unresectable Hepatocellular Carcinoma: Protocol for the STOP-HCC Phase 3 Randomized Controlled Trial. JMIR Res Protoc. 2018 Aug 15;7(8):e11234. doi: 10.2196/11234. PMID 30111528
- See also: Trial-specific website — http://www.theraspheretrials.com/stop-hcc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 526 participants were randomized to either the Control Group (Sorafenib + Standard of Care) or the Treatment Group (TheraSphere + Sorafenib + Standard of Care).
Pre-assignment Details: The Overall Survival (OS) efficacy endpoints analyzed on the modified Intent-To-Treat (mITT) population, comprising 481/526 randomized patients who met eligibility criteria.
Groups:
- Sorafenib + Standard of Care: Control group - Modified Intent-to-Treat (mITT)
- TheraSphere + Sorafenib + Standard of Care: Treatment group - Modified Intent-to-Treat (mITT)
  TheraSphere: Yttrium 90 microspheres
Period: Randomized Patients Summary
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Started (The Overall Survival (OS) efficacy endpoints analyzed on the modified Intent-To-Treat (mITT) population, comprising 481/526 randomized patients who met eligibility criteria.) | 263 | 263
Completed | 241 | 240
Not Completed | 22 | 23
Not completed — Protocol Violation | 22 | 23
Period: Overall Survival (OS)
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Started (Modified Intent-to-treat (mITT) Population: all randomized patients who met the trial eligibility criteria at randomization formed the mITT population. Patients were analyzed according to the group to which they were randomized. This population was used for all efficacy endpoints.) | 241 | 240
Completed (mITT: Patients who died and patients who remained in follow-up at the data cut-off date (30Apr2022), are considered to have completed the study.) | 229 (Treated Patients who Discontinued/Completed from Study) | 222 (Treated Patients who Discontinued/Completed from Study)
Not Completed | 12 | 18
Not completed — Untreated Patients who Discontinued/Completed from Study | 12 | 18

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib + Standard of Care: Control group: Standard-of-care sorafenib, with no added therapy
- TheraSphere + Sorafenib + Standard of Care: Treatment group: Standard-of-care sorafenib plus TheraSphere
  TheraSphere: Yttrium 90 microspheres
- Total: Total of all reporting groups
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care | Total
Number analyzed (Participants) | 241 | 240 | 481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 130 | 120 | 250
  >=65 years | 111 | 120 | 231
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 215 | 210 | 425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 144 | 136 | 280
  Unknown or Not Reported | 91 | 100 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 55 | 52 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 9 | 11
  White | 95 | 79 | 174
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 85 | 97 | 182
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 21 | 43
  South Korea | 47 | 43 | 90
  Belgium | 2 | 1 | 3
  United States | 26 | 34 | 60
  Netherlands | 4 | 4 | 8
  United Kingdom | 28 | 22 | 50
  France | 80 | 94 | 174
  Germany | 1 | 3 | 4
  Spain | 28 | 15 | 43
  Hong Kong | 2 | 0 | 2
  Singapore | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Results Are Based on the Modified Intent-to-treat (mITT)
Description: Time from randomization until date of death due to any cause as reported by study site.
Time Frame: From time of randomization up to date of death or last date known to be alive (data cut-off 30Apr2022), an average of 16.3 months
Population: All participants were analyzed, and the count of participants is reporting the number of events (deaths).
Measure: Count of Participants; unit: Participants
Groups:
- Sorafenib + Standard of Care: Control group - Modified Intent-to-Treat (mITT): Standard-of-care sorafenib, with no added therapy
- TheraSphere + Sorafenib + Standard of Care: Treatment group - Modified Intent-to-Treat (mITT): Standard-of-care sorafenib plus TheraSphere
  TheraSphere: Yttrium 90 microspheres
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 241 | 240
Participants | 200 | 206
Statistical Analysis 1: Comparison: Sorafenib + Standard of Care vs TheraSphere + Sorafenib + Standard of Care; Test type: Superiority; p = 0.4552, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.89 to 1.31]

2. Primary Outcome: Overall Survival (OS) Per Protocol (PP) Population
Description: Per Protocol = subset of the mITT population excluding patients with major protocol deviations which may affect the efficacy evaluation.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sorafenib + Standard of Care: Control group - Per Protocol (PP) Population: Standard-of-care sorafenib, with no added therapy
- TheraSphere + Sorafenib + Standard of Care: Treatment group - Per Protocol (PP) Population: Standard-of-care sorafenib plus TheraSphere
  TheraSphere: Yttrium 90 microspheres
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 218 | 104
Months | 13.2 [11.9 to 14.8] | 13.8 [11.1 to 20.3]
Statistical Analysis 1: Comparison: Sorafenib + Standard of Care vs TheraSphere + Sorafenib + Standard of Care; Test type: Superiority; p = 0.0626, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.61 to 1.01]

3. Secondary Outcome: Time to Progression (TTP) From Time of Randomization Based on Investigator, According RECIST Criteria.
Description: Time to progression (TTP) will be calculated as the interval between the randomization date and the date of first disease progression, including the appearance of new lesion(s) (per RECIST 1.1) and death for any cause or of last contact for patients alive.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 241 | 240
Months | 5.6 [5.5 to 8.0] | 8.1 [6.7 to 11.0]
Statistical Analysis 1: Comparison: Sorafenib + Standard of Care vs TheraSphere + Sorafenib + Standard of Care; Test type: Superiority; p = 0.0227, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [.59 to .96]

4. Secondary Outcome: Time to Untreatable Progression (TTUP) From the Time of Randomization Based One or More of the Following: Investigator Assessment According to RECIST Criteria
Description: Time to progression (TTP) will be calculated as the interval between the randomization date and the date of first disease progression, including the appearance of new lesion(s) and death for any cause or of last contact for patients alive.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 241 | 240
Months | 8.0 [5.6 to 11.2] | 12.2 [9.5 to 16.5]
Statistical Analysis 1: Comparison: Sorafenib + Standard of Care vs TheraSphere + Sorafenib + Standard of Care; Test type: Superiority; p = 0.0043, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [.52 to .89]

5. Secondary Outcome: Tumor Response
Description: Objective Response Rate by investigator determination per RECIST 1.1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 241 | 240
Participants | 20 | 57
Statistical Analysis 1: Comparison: Sorafenib + Standard of Care vs TheraSphere + Sorafenib + Standard of Care; Test type: Superiority; p = 0.0001, 2 sided calculated using continuity; 2 sided calculated using continuity adjusted Wald Approach; Mean Difference (Final Values) = 15.5, 95% CI 2-sided [8.6 to 22.3]

6. Post Hoc Outcome: Summary of Protocol Deviations
Description: A modified Intention To Treat (mITT) Population was used to analyze all efficacy endpoints. This population is defined as randomized patients who met the study eligibility criteria at randomization. This outcome analysis is based on the mITT population, which includes patients with major protocol deviations.
Time Frame: From time of randomization up to date of death or last date known to bealive (data cut-off 30Apr2022), an average of 16.3 months
Population: Percentages are based on the number of patients in each treatment group. A major protocol deviation is a deviation that may affect efficacy evaluation and results in removal of a patient from Per Protocol Population. Of the Major protocol deviations 156/159 patients had treatment related exclusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
Number analyzed (Participants) | 241 | 240
Participants
  Patients with a Major Protocol Deviation | 23 | 136
  Patients with a Protocol Deviation | 193 | 225

ADVERSE EVENTS:
Time Frame: From time of randomization up to date of death or last date known to be alive (data cut-off 30Apr2022), an estimated average of 16.3 months.
Description: Based on patients who received any amount of study treatment. For Control arm patients, AEs were documented for 30 days from the date of discontinuation. After this, only AEs related to TheraSphere were collected. AEs were summarized based on treatment received rather than treatment assigned; therefore, patients at risk is different compared to patients randomized and eligible (miTT). AE summaries include patients that were not in the mITT, therefore, certain events (e.g. deaths) may be higher.
Arm/Group | Sorafenib + Standard of Care | TheraSphere + Sorafenib + Standard of Care
All-Cause Mortality (participants affected / at risk) | 239/274 | 178/207
Serious Adverse Events (participants affected / at risk) | 111/274 | 94/207
Other Adverse Events (participants affected / at risk) | 259/274 | 189/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Standard of Care (N=274) | TheraSphere + Sorafenib + Standard of Care (N=207)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (5) | 10 (12)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (2)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (3)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 13 (13) | 14 (14)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 6 (7) | 5 (5)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Sudden death (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 10 (10) | 10 (11)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (4) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation hepatitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 8 (8)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Posterior reversible encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 4 (4)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Therapeutic embolisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Standard of Care (N=274) | TheraSphere + Sorafenib + Standard of Care (N=207)
Anaemia (Blood and lymphatic system disorders) | 18 (30) | 13 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (19) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 54 (67) | 42 (54)
Abdominal pain upper (Gastrointestinal disorders) | 18 (19) | 12 (13)
Ascites (Gastrointestinal disorders) | 38 (47) | 42 (48)
Constipation (Gastrointestinal disorders) | 36 (37) | 26 (29)
Diarrhoea (Gastrointestinal disorders) | 140 (234) | 62 (92)
Nausea (Gastrointestinal disorders) | 50 (60) | 44 (65)
Stomatitis (Gastrointestinal disorders) | 18 (23) | 8 (8)
Vomiting (Gastrointestinal disorders) | 27 (31) | 26 (33)
Asthenia (General disorders) | 22 (28) | 42 (60)
Fatigue (General disorders) | 84 (128) | 69 (109)
Oedema peripheral (General disorders) | 32 (40) | 26 (32)
Pain (General disorders) | 12 (12) | 15 (15)
Pyrexia (General disorders) | 17 (24) | 23 (23)
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 (10) | 15 (18)
Aspartate aminotransferase increased (Investigations) | 14 (15) | 10 (11)
Blood bilirubin increased (Investigations) | 14 (24) | 22 (26)
Weight decreased (Investigations) | 43 (70) | 30 (37)
Decreased appetite (Metabolism and nutrition disorders) | 87 (130) | 64 (90)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (19) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (9) | 10 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (28) | 14 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (30) | 9 (12)
Headache (Nervous system disorders) | 12 (12) | 11 (13)
Insomnia (Psychiatric disorders) | 6 (6) | 13 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 12 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 12 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 36 (38) | 15 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (16) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (20) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 31 (40) | 18 (26)
Hypertension (Vascular disorders) | 61 (91) | 28 (35)

LIMITATIONS AND CAVEATS:
There were considerably more patients excluded from the TheraSphere arm than the control arm in the per protocol population, this is based on Major Protocol Deviations many of which were related to non-compliance with treatment regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT01556490/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT01556490/SAP_001.pdf